CLINICAL TRIAL: NCT05956795
Title: Surveillance of Regional Nodal Basins in Patients With Primary High Risk Cutaneous Squamous Cell Carcinoma of the Head and Neck
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00270545
Record Dates: First submitted 2023-07-12; First posted 2023-07-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cutaneous Squamous Cell Carcinoma of the Head and Neck
Keywords: ultrasound; Brigham and Women's Hospital Staging; high risk cutaneous squamous cell carcinoma; head and neck; lymph node basins; immunosuppressed; BWH
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- BWH stage T2a tumors in patients who are on chronic immunosuppression: Patient's whose cutaneous squamous cell carcinoma is BWH stage T2a and also have a history of organ transplant, hematologic malignancy, autoimmune disease. After these participants are diagnosed, the participants are entered into the study without any further imaging or sentinel lymph node biopsy. The participants will have ultrasound surveillance every 6 months and regular visits every 3 months throughout the duration of the study (2 years).
  Interventions: Diagnostic Test: Ultrasound
- BWH stage T2b: Participants whose cutaneous squamous cell carcinoma is BWH stage T2b. Participants will initially undergo CT imaging of the nodal basin immediately after diagnosis. If the CT is positive, the participants will be excluded from the study. If the CT is unremarkable, patients will undergo sentinel lymph node biopsy (SLNB), which has a higher sensitivity to detect occult micro-metastases. If the SLNB is negative, the participants are entered into the study. The participants will have ultrasound surveillance every 6 months and regular visits every 3 months throughout the duration of the study (2 years).
  Interventions: Diagnostic Test: Ultrasound
- BWH stage T3: Participants whose cutaneous squamous cell carcinoma is BWH stage T3. Participants will initially undergo CT imaging of the nodal basin immediately after diagnosis. If the CT is positive, The participants will be excluded from the study. If the CT is unremarkable, patients will undergo sentinel lymph node biopsy (SLNB), which has a higher sensitivity to detect occult micro-metastases. If the SLNB is negative, the participants are entered into the study The participants will have ultrasound surveillance every 6 months and regular visits every 3 months throughout the duration of the study (2 years).
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Sonographic imaging will be performed of lymph node basins

SUMMARY:
In this prospective cohort study, investigators will conduct ultrasound surveillance of the nodal basins of patients with head and neck cutaneous squamous cell carcinoma (cSCC) whose tumors are considered high risk and staged by the Brigham and Women's Hospital (BWH) tumor staging system. The study will enroll patients with tumors staged T2a and who are also immunosuppressed (from solid organ transplant, hematologic malignancy or autoimmune disease), T2b (sentinel lymph node negative), and T3 (sentinel lymph node negative). After two years of surveillance, outcomes regarding local recurrence, nodal metastasis, disease specific death, and overall survival will be compared with historical controls with the overall hypothesis that ultrasound surveillance will detect subclinical disease earlier and help improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All cSCC must be on the head or neck
* All cSCC must be primary tumors.
* BWH stage T2a tumors in patients who are on chronic immunosuppression (organ transplant, hematologic malignancy, autoimmune disease)
* All BWH T2b or T3 tumors with a negative CT of the nodal basin AND a negative SLNB

Exclusion Criteria:

* Recurrent tumors
* Patients who are BWH T2b/T3 who have a positive CT of the nodal basin or positive lymph node biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from outpatient general dermatology clinics and surgical clinics in The Johns Hopkins system. Patients who are referred to the The Johns Hopkins system for research purposes will also be considered.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-08-14 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Nodal metastasis | From diagnosis up to 2 years
  Metastatic squamous cell carcinoma to lymph node basins will be assessed through regular US surveillance of each cohort group along with review of respective medical records for any subsequent studies that were performed to confirm metastasis during routine care. Review of medical records will be conducted for historical controls.
  Investigators will then compare time to nodal metastasis between the US surveillance group and the historical controls using Kaplan-Meier estimates of the survivor function and a log-rank test. The investigators will also use Cox proportional-hazards regression to estimate the hazard ratio of nodal metastasis between these two group while adjusting for the covariates of age, sex, stage, etc.

SECONDARY OUTCOMES:
Number of participants with local recurrence of squamous cell carcinoma | From diagnosis up to 2 years
  Recurrent squamous cell carcinoma in the original excision site will be confirmed by review of respective medical records/charts for subsequent confirmation studies performed during routine care.
  Investigators will use Kaplan-Meier estimates, a log-rank test, and Cox proportional-hazards to compare time to local recurrence between groups
Disease specific death | From diagnosis up to 2 years
  Death from cutaneous squamous cell carcinoma will be determined by review of medical records.
  Investigators will compare two-year disease-specific mortality rates between groups using a test of two proportions followed by logistic regression to allow adjustment for covariates.
Overall survival rate | From diagnosis up to 2 years
  The percentage of participants in each cohort who are still alive at the end of the study.
  Investigators will compare two-year overall mortality rates between groups using a test of two proportions followed by logistic regression to allow adjustment for covariates

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bibee, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lukowiak TM, Aizman L, Perz A, Miller CJ, Sobanko JF, Shin TM, Giordano CN, Higgins HW 2nd, Etzkorn JR. Association of Age, Sex, Race, and Geographic Region With Variation of the Ratio of Basal Cell to Cutaneous Squamous Cell Carcinomas in the United States. JAMA Dermatol. 2020 Nov 1;156(11):1192-1198. doi: 10.1001/jamadermatol.2020.2571. PMID 32845319
- [Background] Karia PS, Han J, Schmults CD. Cutaneous squamous cell carcinoma: estimated incidence of disease, nodal metastasis, and deaths from disease in the United States, 2012. J Am Acad Dermatol. 2013 Jun;68(6):957-66. doi: 10.1016/j.jaad.2012.11.037. Epub 2013 Feb 1. PMID 23375456
- [Background] Que SKT, Zwald FO, Schmults CD. Cutaneous squamous cell carcinoma: Incidence, risk factors, diagnosis, and staging. J Am Acad Dermatol. 2018 Feb;78(2):237-247. doi: 10.1016/j.jaad.2017.08.059. PMID 29332704
- [Background] Bander TS, Nehal KS, Lee EH. Cutaneous Squamous Cell Carcinoma: Updates in Staging and Management. Dermatol Clin. 2019 Jul;37(3):241-251. doi: 10.1016/j.det.2019.03.009. PMID 31084718
- [Background] Farasat S, Yu SS, Neel VA, Nehal KS, Lardaro T, Mihm MC, Byrd DR, Balch CM, Califano JA, Chuang AY, Sharfman WH, Shah JP, Nghiem P, Otley CC, Tufaro AP, Johnson TM, Sober AJ, Liegeois NJ. A new American Joint Committee on Cancer staging system for cutaneous squamous cell carcinoma: creation and rationale for inclusion of tumor (T) characteristics. J Am Acad Dermatol. 2011 Jun;64(6):1051-9. doi: 10.1016/j.jaad.2010.08.033. Epub 2011 Jan 20. PMID 21255868
- [Background] Amin MB, Greene FL, Edge SB, Compton CC, Gershenwald JE, Brookland RK, Meyer L, Gress DM, Byrd DR, Winchester DP. The Eighth Edition AJCC Cancer Staging Manual: Continuing to build a bridge from a population-based to a more "personalized" approach to cancer staging. CA Cancer J Clin. 2017 Mar;67(2):93-99. doi: 10.3322/caac.21388. Epub 2017 Jan 17. PMID 28094848
- [Background] Jambusaria-Pahlajani A, Kanetsky PA, Karia PS, Hwang WT, Gelfand JM, Whalen FM, Elenitsas R, Xu X, Schmults CD. Evaluation of AJCC tumor staging for cutaneous squamous cell carcinoma and a proposed alternative tumor staging system. JAMA Dermatol. 2013 Apr;149(4):402-10. doi: 10.1001/jamadermatol.2013.2456. PMID 23325457
- [Background] Ruiz ES, Karia PS, Besaw R, Schmults CD. Performance of the American Joint Committee on Cancer Staging Manual, 8th Edition vs the Brigham and Women's Hospital Tumor Classification System for Cutaneous Squamous Cell Carcinoma. JAMA Dermatol. 2019 Jul 1;155(7):819-825. doi: 10.1001/jamadermatol.2019.0032. PMID 30969315
- [Background] Que SKT, Zwald FO, Schmults CD. Cutaneous squamous cell carcinoma: Management of advanced and high-stage tumors. J Am Acad Dermatol. 2018 Feb;78(2):249-261. doi: 10.1016/j.jaad.2017.08.058. PMID 29332705
- [Background] Ruiz ES, Karia PS, Morgan FC, Schmults CD. The positive impact of radiologic imaging on high-stage cutaneous squamous cell carcinoma management. J Am Acad Dermatol. 2017 Feb;76(2):217-225. doi: 10.1016/j.jaad.2016.08.051. Epub 2016 Oct 1. PMID 27707594
- [Background] de Bondt RB, Nelemans PJ, Hofman PA, Casselman JW, Kremer B, van Engelshoven JM, Beets-Tan RG. Detection of lymph node metastases in head and neck cancer: a meta-analysis comparing US, USgFNAC, CT and MR imaging. Eur J Radiol. 2007 Nov;64(2):266-72. doi: 10.1016/j.ejrad.2007.02.037. Epub 2007 Mar 27. PMID 17391885
- [Background] Fox M, Brown M, Golda N, Goldberg D, Miller C, Pugliano-Mauro M, Schmults C, Shin T, Stasko T, Xu YG, Nehal K; High Risk Squamous Cell Carcinoma Workgroup; Dermatologic Surgery Section of the Association of Professors of Dermatology. Nodal staging of high-risk cutaneous squamous cell carcinoma. J Am Acad Dermatol. 2019 Aug;81(2):548-557. doi: 10.1016/j.jaad.2018.09.006. Epub 2018 Sep 15. PMID 30227190
- [Background] Maher JM, Schmults CD, Murad F, Karia PS, Benson CB, Ruiz ES. Detection of subclinical disease with baseline and surveillance imaging in high-risk cutaneous squamous cell carcinomas. J Am Acad Dermatol. 2020 Apr;82(4):920-926. doi: 10.1016/j.jaad.2019.10.067. Epub 2019 Nov 2. PMID 31689446
- [Background] Tejera-Vaquerizo A, Canueto J, Llombart B, Martorell-Calatayud A, Sanmartin O. Predictive Value of Sentinel Lymph Node Biopsy in Cutaneous Squamous Cell Carcinoma Based on the AJCC-8 and Brigham and Women's Hospital Staging Criteria. Dermatol Surg. 2020 Jul;46(7):857-862. doi: 10.1097/DSS.0000000000002170. PMID 31567487
- [Background] Navarrete-Dechent C, Veness MJ, Droppelmann N, Uribe P. High-risk cutaneous squamous cell carcinoma and the emerging role of sentinel lymph node biopsy: A literature review. J Am Acad Dermatol. 2015 Jul;73(1):127-37. doi: 10.1016/j.jaad.2015.03.039. PMID 26089049
- [Background] Pampena R, Raucci M, Mirra M, Lombardi M, Piana S, Kyrgidis A, Peccerillo F, Paganelli A, Garbarino F, Pellacani G, Longo C. The role of ultrasound examination for early identification of lymph-node metastasis of cutaneous squamous cell carcinoma: results from a single institutional center. Ital J Dermatol Venerol. 2021 Aug;156(4):479-483. doi: 10.23736/S2784-8671.19.06487-3. Epub 2019 Dec 4. PMID 31804052